CLINICAL TRIAL: NCT01384370
Title: Clinical Evaluation of the APTIMA® HPV 16 18/45 Genotype Assay on the TIGRIS® DTS® System in Women With ASC-US Pap Test Results and in Women 30 Years of Age or Older With Negative Pap Test Results Using ThinPrep Pap Test Specimens
Brief Title: APTIMA HPV 16 18/45 Genotype Assay on the TIGRIS DTS System in Women With ASC-US or Negative Pap Test Results
Acronym: AHPV-GT
Status: Completed | Type: Observational
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: HPVGTS-US10-002
Record Dates: First submitted 2011-02-18; First posted 2011-06-29 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Cervical specimens collected in ThinPrep Pap Test vials containing PreservCyt Solution (Hologic, Inc., Marlborough, Massachusetts) with commercially available collection devices (broom-type collection device or cytobrush/spatula combination)* may be tested with the AHPV-GT Assay either pre- or post-Pap processing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AHPV positive and negative subjects

SUMMARY:
In both the ASC-US Study and Adjunct Study populations, the objectives are to:

* evaluate the performance characteristics of the AHPV-GT Assay for detecting cervical disease in women with APTIMA HPV Assay positive results and
* evaluate the ability of the AHPV-GT Assay to detect HPV high-risk types 16, 18, and 45 in women with APTIMA HPV Assay positive results.

DETAILED DESCRIPTION:
The APTIMA HPV 16 18/45 Genotype Assay (AHPV-GT Assay) is an in vitro nucleic acid amplification test for the qualitative detection of E6/E7 viral messenger RNA (mRNA) of human papillomavirus (HPV) types 16, 18 and 45 in cervical specimens from women with positive results in the APTIMA HPV Assay. The AHPV-GT Assay can differentiate between samples positive for HPV 16 from those positive for HPV 18 and/or 45, but does not differentiate between HPV 18-positive samples and HPV 45-positive samples. Cervical specimens collected in ThinPrep Pap Test vials containing PreservCyt Solution (Hologic, Inc., Marlborough, Massachusetts) with commercially available collection devices (broom-type collection device or cytobrush/spatula combination) may be tested with the AHPV-GT Assay either pre- or post-Pap processing. The assay is used with the TIGRIS DTS (TIGRIS) System.

In both the ASC-US Study and Adjunct Study populations, the objectives are to:

* evaluate the performance characteristics of the AHPV-GT Assay for detecting cervical disease in women with APTIMA HPV Assay positive results and
* evaluate the ability of the AHPV-GT Assay to detect HPV high-risk types 16, 18, and 45 in women with APTIMA HPV Assay positive results.

ELIGIBILITY:
Inclusion Criteria:

* • the subject attended a colposcopy visit, and

  * the referral Pap sample had a valid APTIMA HPV Assay result, and

    * the sample had an APTIMA HPV Assay positive result, or
    * the sample had an APTIMA HPV Assay negative result and the subject had a consensus histology result of cervical intraepithelial neoplasia (CIN) grade 2 [CIN2] or more severe (eg, CIN2, CIN grade 3 [CIN3], or cervical cancer; "CIN2+"), or
    * the sample had an APTIMA HPV Assay negative result and the subject had a consensus histology result of normal or CIN grade 1 (<CIN2) and was randomly selected for inclusion. the referral Pap sample had a valid APTIMA HPV Assay result, and
    * the sample had an APTIMA HPV Assay positive result, or
    * the sample had an APTIMA HPV Assay negative result and the subject had a consensus histology result of CIN2+, or
    * the sample had an APTIMA HPV Assay negative result and the subject had a consensus histology result of <CIN2 and was randomly selected for inclusion.

Exclusion Criteria:

* Samples from evaluable subjects meeting the sample inclusion criteria will not be tested with the AHPV-GT Assay if there is insufficient volume for AHPV-GT Assay testing or the sample was deemed unsuitable for testing (eg, stored under unacceptable conditions).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AHPV Assay positive results (~310 from subjects with a consensus histology result of <CIN2 or indeterminate disease status and 70 from subjects with CIN2+)
  * 150 randomly selected AHPV Assay negative samples from subjects with a consensus histology result of <CIN2 and All AHPV Assay negative samples from subjects with CIN2+ (~13 samples)
  * 300 from subjects with a consensus histology result of <CIN2 or indeterminate disease status, 15 from subjects with CIN2+, and 200 from subjects who did not attend the colposcopy visit) Approximately 150 randomly selected APTIMA HPV Assay negative samples from subjects with a consensus histology result of <CIN2 All APTIMA HPV Assay negative samples from subjects with CIN2+ (approximately 5 samples)
Sampling Method: Non-Probability Sample
Enrollment: 1260 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the assay to detect HPV genotypes 16, 18 and/or 45 | 6 months
  Sensitivity (%) = TP/(TP + FN) x 100:
  True Negative (TN): AHPVGT=Negative, Cervical Disease Status <CIN2; True Positive (TP): AHPVGT=Positive, Cervical Disease Status CIN2+; False Positive (FP): AHPVGT=Positive, Cervical Disease Status <CIN2; False Negative (FN): AHPVGT=Negative, Cervical Disease Status CIN2+; Indeterminate: AHPVGT= Invalid, Cervical Disease Status Any; AHPVGT = APTIMA HPV 16 18/45 Genotype Assay
Specificity of the assay to give a positive signal only in HPV 16, 18 and/or 45 positive samples | 6 months
  Specificity (%) = TN/(TN + FP) x100:
  True Negative (TN): AHPVGT=Negative, Cervical Disease Status <CIN2; True Positive (TP): AHPVGT=Positive, Cervical Disease Status CIN2+; False Positive (FP): AHPVGT=Positive, Cervical Disease Status <CIN2; False Negative (FN): AHPVGT=Negative, Cervical Disease Status CIN2+; Indeterminate: AHPVGT= Invalid, Cervical Disease Status Any; AHPVGT = APTIMA HPV 16 18/45 Genotype Assay

CONTACTS AND LOCATIONS:
Overall Officials: Tadd S Lazarus, M.D., Study Director — Gen-Probe, Incorporated
Locations (3):
- United States (3):
  - North Shore LIJ Health System Laboratories, Lake Success, New York
  - Laboratory Corporation of America, Burlington, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio